CLINICAL TRIAL: NCT01557582
Title: Assessment of Right Ventricular Volume Using the Ventripoint Medical System in Patients With Pulmonary Arterial Hypertension
Brief Title: Assessmet of Patients With PAH Right Ventricular Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VentriPoint Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011052
Record Dates: First submitted 2011-08-30; First posted 2012-03-19 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: IPAH; HPAH; APAH CTD; APAH HIV; APAH PoPH; APAH Drugs/Toxins; APAH CHD repaired; APAH CHD unrepaired
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Right ventrical volumn comparison (Other): Single arm study comparing Ventripoint Medical System (VMS) right ventricle volume measurement to gold standard cardiac Magnetic Resonance Imaging (cMRI) measurement in patients with Pulmonary Arterial Hypertension.
  Interventions: Device: Ventripoint Medical System

INTERVENTIONS:
Device: Ventripoint Medical System — The subjects will undergo a 2D echocardiography according to standard of care. An additional 5 - 10 minutes of scanning using VMS transducer attached to the echocardiography system to acquire images for 3-D reconstruction is required.
  Within one day of the VMS image acquisition the subjects will also undergo cMRI according to hospital standards of care plus an additional 5 minutes to capture the PSSS required images.

SUMMARY:
The primary endpoint of this study is the percent difference between the VentriPoint Medical System (VMS) and cMRI for estimating the end diastolic and end systolic right ventricular volumes (RVEDV and RVESV) in subjects with Pulmonary Arterial Hypertension (PAH). The trial will be defined as positive if the mean VMS-cMRI percent difference is <10% and >-10% at a 1-sided 0.025 statistical significance level for RVEDV and for RVESV, with no safety concerns for the VMS procedure.

DETAILED DESCRIPTION:
The objective of this study is: The comparison of the VMS and MRI values for EDV, ESV, and EF using 75 subjects.

Secondary objectives are:

The determination of VMS inter-observer and intra-observer variability of these quantities using 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Group 1 Pulmonary Arterial Hypertension
* IPAH
* HPAH
* APAH-CTD
* APAH-HIV
* APAH-PoPH
* APAH-Drugs/Toxins
* APAH-CHD repaired simple systemic to pulmonary shunts, i.e. ASD, VSD and/or PDA
* APAH-CHD unrepaired simple systemic to pulmonary shunts, i.e. ASD, VSD and/or PDA Patients who can be expected to lie motionless during imagine Males and females 12 years of age and older

Exclusion Criteria:

* Lack of informed consent (and assent as appropriate)
* Other forms of PH not included in inclusion criteria
* Left heart disease including clinically significant valvular disease, ,i.e. moderate or greater mitral regurgitation or stenosis or mild or greater aortic insufficiency or stenosis, pericardial disease, LV systolic dysfunction, i.e. LVEF <40% or LVSF <22%, and/or clinically significant LVDD
* Known/detected arrhythmia that interferes with image acquisition
* Implanted cardiac defibrillator, pacemaker, or other devices containing ferromagnetic materials
* Pregnant or breast-feeding females
* Contraindications for MRI (for those patient that undergo MRI)
* Clinically significant obstructive or restrictive lung disease
* Subjects with known HIV infection who have any clinical or laboratory evidence of any opportunistic pulmonary disease (e.g., tuberculosis, Pneumocystis carinii pneumonia, or other pneumonias)
* PAH associated with thyroid disorders, glycogen storage disease, Gaucher's disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders or splenectomy
* Any subjects with congenital heart disease other than the simple congenital to systemic shunts specified in the inclusion criteria
* PAH associated with significant venous or capillary involvement (PCWP ˃ 15 mmHg), known pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis
* Clinically significant cardiac ischemic disease
* Systemic hypertension defined as SBP ˃ 160 mmHg and/or DBP ˃ 95 mmHg (treated or untreated)
* Moderate or severe hepatic impairment, i.e., Child-Pugh Class B or C
* Any subject with obstructive sleep apnea or who requires the use of CPAP or BiPAP device

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Barst, MD, Principal Investigator — Scientific Advisory Board
Locations (7):
- United States (6):
  - University of Chicago, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baylor, Houston, Texas
- Toronto General Hospital, Tononto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Ventrical Volume Comparison: Single arm study comparing Ventripoint Medical System (VMS) right ventricle volume measurement to gold standard cardiac Magnetic Resonance Imaging (cMRI) measurement in patients with Pulmonary Arterial Hypertension.
  Ventripoint Medical System: The subjects will undergo a 2D echocardiography according to standard of care. An additional 5 - 10 minutes of scanning using VMS transducer attached to the echocardiography system to acquire images for 3-D reconstruction is required.
  Within one day of the VMS image acquisition the subjects will also undergo cMRI according to hospital standards of care plus an additional 5 minutes to capture the PSSS required images.
Period: Overall Study
Arm/Group | Right Ventrical Volume Comparison
Started | 103
Completed | 97
Not Completed | 6
Not completed — Protocol Violation | 4
Not completed — Operator error | 2

BASELINE CHARACTERISTICS:
Population: Demographic information was not available for 2 patients. One subject failed to disclose metal in his abdomen and the other was due to user error.
Arm/Group | Right Ventrical Volume Comparison
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6
  African American | 17
  Native American/Nat. Alaska | 1
  Native Hawaii/Pac Island | 0
  White/Caucasian | 65
  Hispanic/Latino | 12
Region of Enrollment [Number; unit: participants]
  United States | 84
  Canada | 17
WHO Functional Health Class [Number; unit: participants] — The World Health Organization (WHO) has developed a system to help doctors determine how limited a patient is in their ability to do the activities of daily living. In general, patients with more severe PH tend to have a higher functional class.
  Class I: pulmonary hypertension without resulting limitation of physical activity; Class II: slight limitation of physical activity; Class III: marked limitation of physical activity.
  participants
    Functional Class I | 7
    Functional Class II | 46
    Functional Class III | 48
Etiology [Number; unit: participants]
  CONNECTIVE TISSUE | 39
  PORTAL HYPERTENSION | 2
  Simple Congenital | 6
  Drug/Toxin | 4
  Idiopathic | 46
  HIV Infection | 1
  Heritable | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Observed Mean (Std Err) for % Difference Between VMS and MRI.
Description: % Difference was measured for right ventricular EDV, ESV and EF.
Time Frame: VMS occured on day 1 and required 15 minutes and MRI occurred on day 1 and required 1 hour.
Population: Only evaluable participants were analyzed
Measure: Mean (Standard Error); unit: Percent difference
Arm/Group | Right Ventrical Volume Comparison
Number analyzed (Participants) | 75
Percent difference
  EDV | 4.80 (1.35)
  ESV | 1.76 (1.51)
  EF | 2.03 (0.66)
Statistical Analysis 1: Comparison: Right Ventrical Volume Comparison; Test type: Superiority or Other; EDV percent difference = 4.80, 95% CI 2-sided [2.24 to 7.56] — Mean percent difference and 95% CI for EDV
Statistical Analysis 2: Comparison: Right Ventrical Volume Comparison; Test type: Superiority or Other; ESV percent difference = 1.76, 95% CI 2-sided [-1.17 to 4.76] — Mean percent difference and 95% CI for ESV
Statistical Analysis 3: Comparison: Right Ventrical Volume Comparison; Test type: Superiority or Other; EF percent difference = 2.03, 95% CI 2-sided [0.72 to 3.33] — Mean percent difference and 95% CI for EF

2. Secondary Outcome: Inter-Observer Variability
Description: A VMS/echo inter-observer analysis of VMS between-Observer Variation for N=75 Studies.
Time Frame: VMS occured on day 1 and required 15 minutes and MRI occurred on day 1 and required 1 hour.
Population: All evaluable subjects.
Measure: Mean (Standard Deviation); unit: Percent difference
Arm/Group | Right Ventrical Volume Comparison
Number analyzed (Participants) | 75
Percent difference
  EDV Observer 2 vs. 1 | 12.99 (10.59)
  EDV Observer 3 vs. 1 | 18.41 (16.45)
  EDV Observer 3 vs. 2 | 18.49 (15.05)
  ESV Observer 2 vs. 1 | 10.13 (8.60)
  ESV Observer 3 vs. 1 | 15.10 (13.90)
  ESV Observer 3 vs. 2 | 14.38 (12.53)
  EF Observer 2 vs. 1 | 5.83 (4.51)
  EF Observer 3 vs. 1 | 6.12 (5.46)
  EF Observer 3 vs. 2 | 6.83 (5.33)

3. Secondary Outcome: Intra-Observer Variability
Description: Intra-Observer Variation: Directional Difference within Observer (Reading 2-Reading 1)
Time Frame: VMS occured on day 1 and required 15 minutes and MRI occurred on day 1 and required 1 hour.
Measure: Mean (Standard Deviation); unit: Percent difference
Arm/Group | Right Ventrical Volume Comparison
Number analyzed (Participants) | 35
Percent difference
  EDV Observer 1 | 1.41 (6.40)
  EDV Observer 2 | 2.43 (11.92)
  EDV Observer 3 | 3.48 (20.51)
  ESV Observer 1 | 4.01 (4.99)
  ESV Observer 2 | 1.66 (10.32)
  ESV Observer 3 | 10.72 (20.38)
  EF Observer 1 | -1.33 (2.00)
  EF Observer 2 | 0.15 (4.49)
  EF Observer 3 | -3.02 (8.81)

ADVERSE EVENTS:
Time Frame: Adverse events were only collected during imaging.
Arm/Group | Right Ventrical Volume Comparison
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less